CLINICAL TRIAL: NCT06360848
Title: Surgical Treamtment of Pseudarthrosis of the Humerus (Study of a Series of 53 Cases)
Status: Completed | Type: Observational
Sponsor: Ibn Jazzar Hospital (Other)
Responsible Party: Principal Investigator, Zied Mansi, Principal invastigator, Ibn Jazzar Hospital
Other Study IDs: IRB00001192
Record Dates: First submitted 2024-03-26; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Humerus Fracture
Keywords: humerus; pseudarthrosis; screwed plate; external fixator
MeSH Terms: conditions — Humeral Fractures; Pseudarthrosis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: surgery — SURGICAL TREATMENT OF PSEUDARTHROSIS OF THE HUMERUS

SUMMARY:
Pseudarthrosis of the humerus is a serious complication of humerus fractures, of particular interest to subjects young working people with pseudoarthrogenic risk factors (tobacco++). It represents a real problem therapeutic given the long period of treatment, its disabling socio-professional repercussions and the cost which resulting.

The aim of our work is to evaluate the anatomical and functional results of different surgical techniques. used.

DETAILED DESCRIPTION:
The management of pseudarthrosis of the humerus remains a subject of controversy. Given our results, the investigators think that osteosynthesis by plate associated with bone grafting and/or decortication remains the most suitable for the treatment of aseptic pseudarthroses of the humeral shaft while treatment with Ilizarov is most appropriate in septic pseudarthrosis.

However, the best treatment for pseudarthrosis of the humerus remains that of treating the initial fracture. and better control of pseudoarthrogenic risk factors (tobacco++).

ELIGIBILITY:
Inclusion Criteria:

* - Adult men and women > 18 years old with pseudarthrosis of the post-fractured humeral diaphysis treated in the orthopedic surgery and traumatology department.

Exclusion Criteria:

* - Unusable files.
* Patients lost to follow-up.
* Patients who did not accept therapeutic treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 53 cases. of pseudarthrosis of the humeral shaft collected at the surgery department orthopedic and traumatology
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Distribution of atrophic pseudarthrosis according to technique surgical procedure used (in Number of patients) | a minimum follow-up of 10
  Surgical technique Screwed plate:5 Percutaneous pinning:12
Distribution of hypertrophic pseudarthrosis according to technique surgical procedure used (in Number of patients) | a minimum follow-up of 10 months
  Surgical technique Screwed plate:4 Percutaneous pinning:9
Time to consolidation depending on the type of pseudarthrosis (in months) | a minimum follow-up of 10 months
  Atrophic Pseudarthrosis 4.4 months Pseudarthrosis Aseptic 5.28 months Hypertrophic Pseudarthrosis 5.8 months Septic Pseudarthrosis 4.6 months
Average Constant score postoperatively according to the means of restraint | a minimum follow-up of 10 months
  Screwed plate(24) :74 External fixator(28) :64 Nailing centromedullary(1) :69

IPD SHARING:
Plan to Share IPD: No